CLINICAL TRIAL: NCT06042231
Title: Impact of Cardiac Prehabilitation, REhabilitation and Patient EDucation on Outcomes in Patients Undergoing First-time AF Ablation
Acronym: CREED AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FO596122
Record Dates: First submitted 2023-08-21; First posted 2023-09-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation
Keywords: AF ablation; Pulmonary vein isolation; VO2peak
MeSH Terms: conditions — Atrial Fibrillation | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental)
  Interventions: Behavioral: Exercise Intervention; Behavioral: Education Intervention
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise Intervention — Exercise and education intervention. Participants will be prescribed a tailored exercise program to complete before ('pre-habilitation') and after their AF ablation procedure (rehabilitation).
  Arms: Exercise Intervention
Behavioral: Education Intervention — Education intervention. Participants will be given a 1-1 education session (up to 3 sessions) before and after their AF ablation procedure. Participants will be given behavioural strategies to improve adherence and compliancec to risk-factor modification.
  Arms: Exercise Intervention

SUMMARY:
Atrial fibrillation (AF) is a term used to describe an irregular, and often very rapid, heartbeat. AF increases the risk of a number of diseases associated with the heart and cardiovascular system. Ablation is a procedure to treat AF. It uses small burns or freezes to cause some scarring on the inside of the heart to help break up the electrical signals that cause irregular heartbeats. This can help the heart maintain a normal rhythm.

Currently patients who are referred for AF ablation do not receive any additional support as part of standard care to improve the outcomes of their ablation procedure. Whereas cardiac rehabilitation is a recognised part of comprehensive care for coronary heart disease patients (patients whose hearts struggle to receive blood), with exercise and education consistently identified as central elements to their rehabilitation. This treatment is not yet recommended for AF ablation patients.

Therefore, the CREED AF Study is investigating whether a tailored comprehensive exercise and education intervention can improve outcomes in patients who are undergoing first time AF ablation. Central to the CREED AF study is the 'prehabilitation' intervention, whereby exercise and education training will be conducted before AND after AF ablation. 106 participants is the target recruitment, they will be randomised to either receive the CREED AF intervention (exercise and education intervention before AND after AF ablation) or a standard care (control) group. The standard care group will receive a one off 1-to-1 patient education session with a trained practitioner before their AF ablation procedure. This research study does not affect the AF ablation procedure that patients will have as part of their standard of care.

DETAILED DESCRIPTION:
This is a single centre, prospective, randomised controlled trial. The CREED AF study will run from University Hospitals Coventry & Warwickshire (UHCW) NHS Trust. There will be collaboration with Atrium Health, a non-profit exercise rehabilitation centre located in Coventry, UK. Atrium Health was founded by frontline NHS clinical staff to provide people with tailored exercise and education programmes. Patients with AF who are referred for first-time AF ablation at University Hospitals Coventry & Warwickshire NHS Trust will be recruited to the trial. The aim is to explore the effectiveness of a tailored comprehensive cardiac rehabilitation programme (both before and after the planned AF ablation) comprising of an exercise programme and patient education programme incorporating lifestyle behaviour change (CREED AF intervention), compared to standard care (control arm).

The CREED AF intervention will involve a cardiac pre/rehabilitation exercise training programme combined with a patient education programme.

To ensure generalisability for future trials, provisions will be based on current delivery models of cardiac rehabilitation in cardiovascular diseases. A 6-8-week supported programme of 2-3 times weekly exercise will be delivered with an initial individual assessment for each patient randomised to the intervention. Participants will attend a one-to-one appointment with a 'CREED AF practitioner' (specialist cardio-pulmonary clinical exercise physiologist or physiotherapist) for the assessment of medical history, medication, clinical parameters, physical activity history and discussion of participant goals, expectations, fears, and concerns. Patients randomised to the CREED AF intervention will have access to both existing cardio-pulmonary rehabilitation programmes at the Atrium Health Centre, Coventry (i.e., they will exercise alongside people with a range of cardio-pulmonary disorders at already running sessions) AND instructor-led, at home workout sessions that will take place live over a video conferencing software. It is anticipated that participants randomised to the CREED AF intervention will choose to receive a hybrid of the two approaches to reduce travel constraints of getting to and from the Atrium Health Centre, and to work more flexibly around a participant's working/personal life. To maximise accessibility and resource, whilst ensuring benefits are retained, the CREED AF intervention will be delivered as a 'rolling' programme. Participants randomised to the CREED AF intervention can immediately join existing cardio-pulmonary rehabilitation exercise programmes rather than waiting for the recruitment of sufficient numbers to form a discrete group of trial participants.

Cardiac pre/rehabilitation This will be a tailored, individualised exercise programme within pre-specified parameters. Clinical information, data from the exercise assessment, and patient-centred goal setting will be used to devise a safe and effective exercise prescription which can be performed either using pre-existing cardiopulmonary exercise groups at Atrium Health or using the instructor-led online classes that will be available. Exercise guidance, specific to AF, will be delivered on an individual basis during a 1-to-1 familiarisation exercise session in the first week of the programme, and reinforced throughout, by clinical staff. Familiarisation sessions, conducted within the cardiopulmonary rehabilitation programmes will enable participants to build their confidence and there will be optimisation of the exercise prescribed.

The cardiac rehabilitation can be undertaken within existing cardio-pulmonary rehabilitation programmes delivered by NHS clinical staff. Up to 3 times weekly, one hour, exercise sessions for 6-8 weeks before and for 6-8 weeks after AF ablation, with a quantifiable and progressive dose of individualised, multi-modal, aerobic, muscular strength, endurance and 'functional fitness' exercise. Adequate warm-up and cool-down will be incorporated. Intensity can be monitored and adjusted using heart rate (where appropriate), rating of perceived exertion, and dyspnoea scale. There is normally a 1-2-week recovery period after an AF ablation procedure to allow for femoral access site wound healing. Only after the participant has completed this 2-week recovery period will they restart their exercise intervention.

The exercise component will be optimised to be appropriate for a broad spectrum of patients including frailer, deconditioned, low-mobility, exercise-naive participants. Conventional gym exercise will be combined with 'functional fitness' training. The programme will be highly adaptable to allow personalisation to lower or higher ability participants, whilst ensuring safety and efficacy. This is widespread practice within cardio-pulmonary rehabilitation programmes in the UK.

In addition to treadmills, cycles, and rowing ergometers, readily available functional fitness equipment such as steps, floor agility ladders, low rise balance beams, power bags, plyometric boxes, balls (throw/bounce) etc will be made use of. A range of body weight exercises for online sessions at home will also be utilised. Central to our intervention is the expertise and experience of the specialist CREED AF practitioner who will ensure holistic, safe, individualised, and effective exercise training.

Education, behavioural and lifestyle AF risk Factor Modification Support The education programme will be delivered in 1-to-1 sessions with a delegated and qualified member of the research team which can be delivered either face-to-face or via an online video conferencing software. The education session will be delivered as part of the CREED AF intervention. Changing behaviours can be difficult and the importance of psychological support in AF patients is recognised. Therefore, discussions with individuals on motivation to change, barriers to change, goal setting and problem-solving to build self-efficacy and encourage behaviour change, adherence, and compliance to risk factor modification will be incorporated. Every second week (a total of 6 1-to-1 education sessions, 3 sessions in prehabilitation before ablation, and 3 sessions in rehabilitation after ablation), before or after exercise, participants will receive a 1-to-1 30-minute behavioural and motivational session with the aim of improving short- and long-term adherence to exercise and lifestyle modification goals. The aim of this will be to provide help to patients to manage lifestyle risk factors. These will include reduction of alcohol consumption to less than 2 Units per day (in line with current UK government guidelines), ensure good blood pressure control in line with international guidelines (<140/85mmHg), provide smoking cessation support, help with good diabetes control, advice on weight reduction management (through diet and exercise) and identification and treatment of obstructive sleep apnoea (OSA). Patients in the intervention group will be provided with written materials, including but not limited to a patient workbook and publicly available patient information leaflets, with sign-posting to support groups as applicable to each individual.

The CPET will be performed by both the control and intervention groups at baseline and 10 weeks (±2 weeks) post-ablation. The test will be used to assess exercise capacity and will give an indicator of the participant's cardiorespiratory fitness. The tests will be performed at UHCW's respiratory laboratory. The lab is UKAS accredited to IQIPS standard to perform CPET. The local UHCW standard operating procedure for CPET will be followed for all participants during their VO2peak test. This information is available in full detail in a separate document, but briefly:

1. The participant will have their height and weight measured and information about the current medications collected.
2. They will have the procedure explained to them in full detail and any questions they have will be answered.
3. A spirometry measurement of forced vital capacity will be obtained before the CPET begins.
4. A 12-lead ECG will be attached to the participant.
5. A Hans Rudolph face mask will be fitted to the participant and baseline data collected.
6. A blood pressure cuff and pulse oximeter will be attached with measurements taken at baseline and during the test.
7. The exercise protocol will begin with increasing exercise intensity until the participant feels they cannot continue, when cadence falls by 5% or more or when the individual leading the exercise test requests it to be stopped.
8. Recovery period involving low intensity exercise.

Participants who are randomised into the control group will also receive a 30-minute 1-to-1 education session (remotely or in person) from a CREED AF practitioner before their AF ablation to go through the risk factors of AF and what they can do to improve their health. The session will involve a discussion with the participant around risk factors related to AF and recommendations for what actions the participant should take to minimise these factors, sign-posting to publicly available patient information leaflets (e.g. https://heartrhythmalliance.org/aa/uk/resources/arrhythmia-alliance-patient-resources). For the rest of the trial, they will follow the standard care pathway for ablation patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients listed for a first-time AF ablation procedure
* Patients aged ≥18 years

Exclusion Criteria:

* Pregnancy
* Lack of capacity to consent and participate
* Presence of contraindications or limiting physical or mental health co-morbidity preventing travel, safe exercise, or productive engagement with the trial
* Unable to access online exercise and support sessions from home
* Participating in a research trial that will impact on their standard AF ablation procedure
* Unable to understand basic spoken and written English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
VO2 peak measurements | 12 months
  VO2peak measured from cardiopulmonary exercise testing (CPET) at baseline and 10 weeks (±2 weeks) post AF ablation between the standard care and intervention arms.

SECONDARY OUTCOMES:
Quality of life questionnaire | 12 months
  EQ-5D-5L questionnaire
Quality of life questionnaire | 12 months
  SF-36 QoL Scale
Quality of life questionnaire | 12 months
  Atrial Fibrillation Effect on Quality-of-Life (AFEQT)
Cost effectiveness of CREED AF intervention | 12 months
  Incremental cost per quality adjusted life year (QALY).
AF recurrence in short- and long-term | 12 months
  AF recurrence and burden from data collected from a 1-7-day(s) cardiac Holter monitoring at 10 weeks (±2 weeks) and 12 months (±4 weeks) post ablation, and requirement for redo-AF ablation as documented in medical records reviewed at 12 months post-ablation.
Occurence of Major Adverse Cardiovascular Events (MACE) | 12 months
  MACE recorded at 12 months post-ablation

CONTACTS AND LOCATIONS:
Overall Officials: Faizel Osman, Principal Investigator — University Hospitals Coventry & Warwickshre NHS Trust
Locations (1):
- University Hospital Coventry and Warwickshire NHS Trust, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Derived] Chandan N, Matthews V, He H, Lachlan T, Lim VG, Joshi S, Hee SW, Noufaily A, Parkes E, Patel S, Andronis L, Shakespeare J, Eftekhari H, Ali A, McGregor G, Osman F. Cardiac prehabilitation, rehabilitation and education in first-time atrial fibrillation (AF) ablation (CREED AF): Study protocol for a randomised controlled trial. PLoS One. 2024 Oct 3;19(10):e0310951. doi: 10.1371/journal.pone.0310951. eCollection 2024. PMID 39361572